CLINICAL TRIAL: NCT02439333
Title: Prospective Randomized Study of Nasal High Flow in Treatment of Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Li Xuyan (Other)
Responsible Party: Sponsor-Investigator, Li Xuyan, Sponsor-Investigator, Beijing Chao Yang Hospital
Organization: Beijing Chao Yang Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-KE-63
Record Dates: First submitted 2015-05-07; First posted 2015-05-08 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2018-05

CONDITIONS: Lung Diseases, Obstructive
Keywords: Acute exacerbation of chronic obstructive pulmonary disease; Nasal high flow therapy; Oxygen therapy
MeSH Terms: conditions — Lung Diseases, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nasal high flow therapy (Active Comparator): AECOPD patients with no severe respiratory insufficiency are given NHF therapy for at least 15 hours per day.
  Interventions: Device: Nasal high flow cannula (Fisher & Paykel Healthcare, Auckland, New Zealand)
- Conventional oxygen therapy (Active Comparator): AECOPD patients with no severe respiratory insufficiency are given conventional oxygen therapy such as nasal catheter or venturi mask for at least 15 hours per day.
  Interventions: Device: nasal catheter or Venturi mask

INTERVENTIONS:
Device: Nasal high flow cannula (Fisher & Paykel Healthcare, Auckland, New Zealand) — Nasal high flow therapy
  Arms: Nasal high flow therapy
Device: nasal catheter or Venturi mask — Conventional oxygen therapy
  Arms: Conventional oxygen therapy

SUMMARY:
The main oxygen therapy to the patients with acute exacerbation of Chronic obstructive pulmonary disease, who are mild to moderate respiratory insufficiency (arterial blood gas analysis showed pH = 7.35, PO2 < 60mmHg,PaCO2>45mmHg) or have achieved the traditional noninvasive ventilation support standard but can not tolerate or reject, was nasal catheter, venturi mask and other conventional oxygen therapy. All these inaccurate inhaled oxygen concentration methods with inadequate heating and humidifying lead to poor patient tolerance and adverse reactions such as airway secretions discharge disorders. The high flow nasal respiratory therapy (Nasal high flow, NHF) utilises higher gas flow rates than conventional low-flow oxygen systems. The devices used deliver heated and humidified oxygen at a flow of up to 60 litres per minute via nasal cannulas with low level continous positive airway pressure. This study is a prospective randomized study. AECOPD patients with no severe respiratory failure are treated with NHF and conventional oxygen therapy respectively. The target is that NHF can increase the comfort degree of patients,reduce the rate of endotracheal intubation, and shorten the time of hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* AECOPD patients.
* The results of blood gas analysis showed pH ≥7.35, PO2< 60mmHg, PaCO2> 45mmHg.

Exclusion Criteria:

* The study case has been incorporated into the hospital again.
* Refused to the NHF therapy.
* The Glasgow score < 8.
* Severe organ dysfunction (including liver and kidney dysfunction, decompensated acidosis, upper gastrointestinal bleeding, DIC, etc.)

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2015-07; Primary Completion 2019-07 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
Treatment failure criteria | 5 days
  Patients with mild respiratory acidosis (7.25 < pH < 7.35) with obvious dyspnea (accessory respiratory muscle involvement, breathing rate greater than 25 beats per minute)

SECONDARY OUTCOMES:
Length of hospital stay | 30 days
Costs of hospitalization expenses | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Bing Sun, MD, Principal Investigator — Beijing Chao Yang Hospital
Locations (1):
- Department of respiratory and critical care medicine,Beijing Chao-yang Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Li XY, Tang X, Wang R, Yuan X, Zhao Y, Wang L, Li HC, Chu HW, Li J, Mao WP, Wang YJ, Tian ZH, Liu JH, Luo Q, Sun B, Tong ZH. High-Flow Nasal Cannula for Chronic Obstructive Pulmonary Disease with Acute Compensated Hypercapnic Respiratory Failure: A Randomized, Controlled Trial. Int J Chron Obstruct Pulmon Dis. 2020 Nov 24;15:3051-3061. doi: 10.2147/COPD.S283020. eCollection 2020. PMID 33262584